CLINICAL TRIAL: NCT05736198
Title: Comparison of Two Sedation Regimens for Awake Fiberoptic Intubation
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, David Glick, Department of Anesthesiology Head, University of Illinois at Chicago
Other Study IDs: 2023-0181
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Awake Fiberoptic Intubation; Difficult Airway
Keywords: Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Dexmedetomidine: Dexmedetomidine, midazolam, and fentanyl (titrated to effect) to facilitate intubation
  Interventions: Drug: Dexmedetomidine
- Placebo: Normal Saline, midazolam, and fentanyl (titrated to effect) to facilitate the intubation

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine, midazolam, and fentanyl (titrated to effect) to facilitate intubation
  Other Names: Precedex
  Groups: Dexmedetomidine

SUMMARY:
The purpose of this study is to examine the effects of different sedation drugs used for the awake fiberoptic intubation procedure. Benzodiazapines and narcotics (such as midazolam and fentanyl) are standard drugs used for sedation during awake fiberoptic intubation. Dexmedetomidine, midazolam, and fentanyl are approved by the Food and Drug Administration (FDA) procedural sedation. These drugs might be given to the patient regardless of their participation in the study.

In addition to midazolam and fentanyl study subjects will also receive either dexmedetomidine or a placebo (a salt solution that contains no drug). It is believed that dexmedetomidine will not slow down breathing as much as the combination of the valium-like drug and narcotic. In our study, we are trying to determine if this is the best drug for sedation during an awake fiberoptic procedure.

DETAILED DESCRIPTION:
This is an observational study designed to evaluate effectiveness of two standard of care protocols used for patients with potentially difficult airway during awake fiberoptic intubation.

After obtaining informed consent, patients will be randomized into one of two groups. The first group will receive placebo, midazolam, and fentanyl (titrated to effect) to facilitate the intubation. The second group will receive dexmedetomidine, midazolam, and fentanyl (titrated to effect) to facilitate intubation. Both groups will have a transtracheal injection and/or direct topical application of lidocaine to decrease irritation of the trachea and vocal cords.

As the patients in the study all have potentially difficult airways, the usual precautions will be taken to minimize the risks to the patients. These include the availability of alternative airway devices (including LMAs and Intubating LMA systems). Doses of dexmedetomidine will conform to the recommended dosing schedules of between 0.3 and 0.7 mcg/kg/hour.

All the drug stated above are currently FDA approved and are used according to the standard of care.

Patient medical records will be reviewed to determine the amount of fentanyl that was used to facilitate intubation as well as homodynamic stability during the procedure and oxygen saturation. A brief 5-minute survey will be conducted 24 hours after the surgery to access patient satisfaction with intubation procedure. Intubation conditions stated below will be recorded by the anesthesiologist during the procedure.

The intubating conditions (gagging, discomfort of patient, and oxygen saturation) and hemodynamic stability during the procedure will be recorded by the research assistant and the patient's satisfaction with the undertaking (after the surgery is completed) will be determined as well. The amount of fentanyl used to facilitate intubation will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with potentially difficult airways who require awake fiberoptic intubations will be identified from the OR schedule and the pre-operative clinic workups.

Exclusion Criteria:

* Anyone who does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults with potentially difficult airways undergoing elective procedures will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2033-06-15 (Estimated); Study Completion 2034-03-01 (Estimated)

PRIMARY OUTCOMES:
Desaturation | During intubation
  Measurement using pulse oximetry (percent saturation)
Hemodynamic Lability | During intubation
  mm Hg
Dose of Fentanyl Used | During intubation
  mcg

SECONDARY OUTCOMES:
Patient overall experience assessed by VAS satisfaction. | 24 hours after the surgery
  Polling will be taken to measure patients' satisfaction with each sedation regiment on the scale from 1-10

CONTACTS AND LOCATIONS:
Overall Officials: David Glick, MD, Principal Investigator — Department of Anesthesiology Head
Locations (1):
- University of Illinois, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Data will only be shared with study investigators

REFERENCES:
- [Background] Scher CS, Gitlin MC. Dexmedetomidine and low-dose ketamine provide adequate sedation for awake fibreoptic intubation. Can J Anaesth. 2003 Jun-Jul;50(6):607-10. doi: 10.1007/BF03018650. PMID 12826556